CLINICAL TRIAL: NCT03700606
Title: Physiological Changes With High-Flow Nasal Cannula Compared to Nasal CPAP in Extremely Low Birth Weight Infants
Brief Title: Physiological Changes With High-Flow Nasal Cannula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director Neonatal Research Institute, Sharp HealthCare
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: HFNC
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Respiratory Distress Syndrome in Premature Infant
Keywords: high flow nasal cannula; nasal cpap

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nasal CPAP - Period 1 (Active Comparator): Eligible infants stable on high flow nasal cannula (nCPAP) therapy of 5-7 cm H20 achieved with a ventilator, an underwater "bubble" system, or a variable-flow device will be enrolled. A data acquisition cart will be placed at the subject's bedside to collect hemodynamic and respiratory parameters measured including: Heart rate (HR), blood pressure (BP), respiratory rate (RR), fraction of inspired oxygen (FiO2), transcutaneous carbon dioxide (TcCO2), and peripheral oxygen saturation (SpO2) via bedside monitoring devices. A neonatal chest belt, sized to the infant's chest circumference (nipple level) using warmed ultrasound gel applied to the belt beforehand, will collect regional lung volume measurements using electrical impedance tomography (EIT). Subject video recording will capture apnea events and the interventions used to resolve them such as positive pressure ventilation, repositioning, or stimulation. Data will be collected for 15 minutes on nCPAP.
  Interventions: Procedure: Nasal CPAP
- High Flow Nasal Cannula (HFNC) - Period 2 & 3 (Active Comparator): Respiratory support will be crossed over to a HFNC Optiflow Jr 2 (Fisher & Paykel Healthcare, Auckland, New Zealand) at a flow rate of 8 LPM. The size of the nasal cannula will be determined according to the manufacturer's instructions in order to maintain a leak at the nares. Identical data collection will occur for two 15 minute periods on HFNC, at the beginning and end of the six hour Study period.
  Interventions: Procedure: High flow nasal cannula
- Nasal CPAP - Period 4 (Active Comparator): After 6 hours of HFNC of 8 LPM, or sooner if the infant meets failure criteria, the infant will then be crossed back to the nCPAP device and at the settings previously utilized in Study Period 1. The infant will remain on the nCPAP device with identical data collection for 15 minutes. The total duration of the study and data collection will be 8 hours. The infant's body position will be similar for each lung volume measurement during the study periods.
  Interventions: Procedure: Nasal CPAP

INTERVENTIONS:
Procedure: High flow nasal cannula — 8 liters per minute of blended oxygen through Fisher Paykel Optiflow Jr 2 nasal prongs.
  Arms: High Flow Nasal Cannula (HFNC) - Period 2 & 3
Procedure: Nasal CPAP — Nasal continuous positive airway pressure of 5-7 cm/H20 delivered using Ventilator or bubble cpap device through short nasal prongs or a nasal face mask.
  Arms: Nasal CPAP - Period 1; Nasal CPAP - Period 4

SUMMARY:
To measure changes in physiologic parameters in extremely low birthweight (ELBW) infants on high-flow nasal cannula compared to nasal continuous positive airway pressure (nCPAP).

DETAILED DESCRIPTION:
After informed consent is obtained, eligible infants who are stable on nCPAP therapy of 5-7 cm H20 achieved with a ventilator, an underwater "bubble" system, or a variable-flow device will be enrolled.

All subjects will have physiologic data and electrical impedance tomography collected at:

1. Baseline nCPAP for 15 minutes
2. Upon transition to high flow nasal cannula at 8 LPM for 6 hours. Data collection is obtained after infant is calm for 15 minutes at the beginning and end of this 6 hour period
3. Then upon return to baseline NCPAP for a final 15 minutes of data collection.

ELIGIBILITY:
Inclusion Criteria:

* 23 to 28+6 weeks gestational age at birth
* Corrected gestational age less than or equal to 30 weeks
* Over 72 hours of life
* Stable on Nasal CPAP of 5-7cm H20
* Hemodynamically stable
* Tolerating routine handling
* Nares size appropriate for Fisher & Paykel Optiflow Jr 2 HFNC size XS or small
* Successfully extubated for 12 hours after administration of surfactant
* Caffeine Citrate at a maintenance dose of 5 to 10 mg /kg
* Transcutaneous monitoring in place
* Stable blood gas (pH>/= 7.25 and PaCO2 <60 mmHg torr)

Exclusion Criteria:

* Prior pneumothorax or evidence of pulmonary interstitial emphysema.
* Prior or current pulmonary hemorrhage
* Congenital airway malformations
* Major cardiopulmonary malformations
* Congenital Diaphragmatic hernia or untreated bowel obstruction
* Poor respiratory drive unresponsive to CPAP therapy
* Requirement of a nCPAP of >8 cmH20 or FiO2 > 0.3 to maintain oxygen saturations between 90-95 percent.
* Receiving positive pressure breaths or SIPAP on prongs
* Conflicting clinical trial
* Clinically unstable per physician discretion

Ages: 23 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
% Unventilated Lung | Through study completion, an average of 30 days
  Atelectasis will be calculated using the percentage of the lung fields that are not engaged in tidal volume.(VT)

SECONDARY OUTCOMES:
Geometric Center of Ventilation (CoV) | Through study completion, an average of 30 days
  numeric value that describes the geographic point within the thorax that represents the statistical center of VT
End-expiratory lung volume | Through study completion, an average of 30 days
  % of total VT within 8 lung regions, relative change in uncalibrated aeration

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Mary Birch Hospital for Women & Newborns, San Diego, California, United States

REFERENCES:
- [Derived] Katheria A, Ines F, Hough J, Rich W, Morales A, Sanjay S, Poeltler D, Finer N. Changes in lung aeration with high-flow nasal cannula compared to nasal CPAP in preterm infants. J Perinatol. 2025 Jun;45(6):817-822. doi: 10.1038/s41372-025-02267-4. Epub 2025 Mar 23. PMID 40122991